CLINICAL TRIAL: NCT04145011
Title: A Prospective, Multi-center, Randomized, Single Blind Clinical Trial Comparing COOLIEF* Cooled Radiofrequency to Conventional Radiofrequency Ablation of the Genicular Nerves in the Management of Knee Pain in an Osteoarthritic Patient Population
Brief Title: Coolief Cooled Radiofrequency vs. Conventional Radiofrequency to Manage OA Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avanos Medical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 105-18-0002
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Osteoarthritis of the Knee
Keywords: Randomized clinical trial; Osteoarthritis; Radiofrequency Ablation; Knee; Genicular; Coolief
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Masking Description: The study is a participant-blinded trial and deliberate action, utilizing a physical barrier, will be needed to ensure the blind remains intact.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- COOLIEF Cooled Radiofrequency Probe (Experimental): Cooled radiofrequency energy will be delivered to the study subjects' knee to ablate culprit sensory nerves and reduce knee pain
  Interventions: Device: Cooled Radiofrequency
- Conventional (Standard) Radiofrequency Probe (Active Comparator): Standard (non-cooled) radiofrequency energy will be delivered to the study subjects' knee to ablate culprit sensory nerves and reduce knee pain
  Interventions: Device: Standard Radiofrequency

INTERVENTIONS:
Device: Cooled Radiofrequency — Delivery of energy to ablate sensory nerves via cooled radiofrequency probe (18g, 4mm active tip)
  Other Names: Coolief, CRFA
  Arms: COOLIEF Cooled Radiofrequency Probe
Device: Standard Radiofrequency — Delivery of energy to ablate sensory nerves via non-cooled standard radiofrequency probe (22g, curved 10mm active tip)
  Other Names: Conventional Radiofrequency, SRFA
  Arms: Conventional (Standard) Radiofrequency Probe

SUMMARY:
This study is being performed to assess the relative effectiveness of genicular nerve ablation with the COOLIEF* Cooled Radiofrequency probe to manage moderate to severe knee pain in patients with osteoarthritis (OA) of the knee when compared to radiofrequency ablation using a Standard Radiofrequency probe.

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized, single-blind comparison study examining the outcomes of subjects with osteoarthritic knee pain undergoing a procedure to create a radiofrequency lesion of the genicular nerves with either Cooled Radiofrequency Ablation (CRFA) or Conventional (Standard) Radiofrequency Ablation (SRFA). Approximately 148 participants from up to 15 sites will be enrolled into this study, with subjects undergoing either CRFA or SRFA in a 1:1 randomization scheme. Follow-up will be conducted for 24 months post-treatment, with the primary endpoint being completed at month 12. Pain, overall outcome, quality of life, pain medication use, and adverse events will be compared between the two treatment groups to determine success.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21 years
2. Able to understand and personally sign and date the informed consent form
3. Able to complete outcome measures
4. Chronic knee pain for longer than 6 months that interferes with functional activities (for example, ambulation, prolonged standing, etc.)
5. Continued pain in the target knee despite at least 3 months of conservative treatments, including activity modification, home exercise, protective weight bearing, and/or analgesics (for example, acetaminophen or non-steroidal anti-inflammatory drugs [NSAIDs])
6. Positive response (defined as a decrease in numeric pain scores of at least 50%) to a single genicular nerve block of the index knee
7. Pain on NRS ≥ 6 on an 11-point scale for the index knee
8. Radiologic confirmation of osteoarthritis (x-ray/MRI/CT) grade 2 (mild), 3 (moderate) or 4 (severe) noted within 6 months for the index knee
9. Analgesics including membrane stabilizers such as Neurontin (gabapentin) and antidepressants for pain, such as Cymbalta (duloxetine), must be clinically stable (defined as stable dosage for ≥ 6 weeks prior to the screening visit) and shall not change during the course of the study without approval of the investigator
10. Agree to see one physician (study physician) for knee pain during the study period
11. Subjects of child bearing potential must be willing to utilize double barrier contraceptive method
12. Willingness to comply with the requirements of this protocol for the full duration of the study (24 months regardless of effect of initial therapy)

Exclusion Criteria:

1. Evidence of inflammatory arthritis (example, rheumatoid arthritis) or other systemic inflammatory condition (example; gout, fibromyalgia, MS, Lupus, etc.) that could cause knee pain
2. Evidence of neuropathic pain affecting the index knee
3. Previous or pending lower limb amputation
4. Intra-articular steroid injection into the index knee within 90 days from randomization
5. Hyaluronic acid injection, platelet rich plasma (PRP), stem cell, or arthroscopic debridement/lavage injection into the index knee within 180 days from randomization
6. Prior radiofrequency ablation of the genicular nerves of the index knee
7. Prior partial, resurfacing, or total knee arthroplasty of the index knee (residual hardware)
8. Clinically significant ligamentous laxity of the index knee
9. Clinically significant valgus/varus deformities or evidence of pathology (other than osteoarthritis of knee) that materially affects gait or function of the knee or is the underlying cause of the knee pain and/or functional limitations
10. Body mass index (BMI) > 40 kg/m2
11. Extremely thin patients and those with minimal subcutaneous tissue thickness that would not accommodate a radiofrequency lesion of up to 14 mm in diameter to limit the risk of skin burns
12. Pending or active compensation claim, litigation, or disability remuneration (secondary gain)
13. Pregnant, nursing or intent of becoming pregnant during the study period
14. Chronic pain associated with significant psychosocial dysfunction
15. Poorly controlled severe psychiatric illness or ongoing psychological barriers to recovery, as determined by the investigator
16. Allergies to any of the medications to be used during the procedures
17. Active joint infection or systemic or localized infection at needle entry sites (subject may be considered for inclusion once infection is resolved)
18. History of uncontrolled coagulopathy, ongoing coagulation treatment that cannot be safely interrupted for procedure, or unexplained or uncontrollable bleeding that is uncorrectable
19. Identifiable anatomical variability that would materially alter the procedure as described in the protocol
20. Within the preceding 2 years, subject has suffered from active narcotic addiction, substance, or alcohol abuse
21. Current prescribed opioid medications greater than 60 mg morphine equivalent daily opioid dose
22. Uncontrolled immunosuppression (e.g. AIDS, cancer, diabetes, etc.)
23. Subject currently implanted with pacemaker, stimulator or defibrillator
24. Participating in another clinical trial/investigation which included therapeutic treatment within 30 days prior to signing informed consent
25. Subject unwilling or unable to comply with follow up schedule, protocol requirements or procedures

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | 12 months
  The proportion of subjects whose knee pain is reduced by ≥ 50% based on the NRS. The NRS is an 11-point scale (0 points to 10 points), where 0 points equals "no pain" and 10 points equals "worst pain". There are no sub-scales.

SECONDARY OUTCOMES:
Additional Interventions | 12 months
  The proportion of subjects requiring additional intervention for their OA knee pain.
Knee injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR) | 12 months
  The change in KOOS JR score from baseline. The KOOS JR is a short form of the KOOS that assesses patient stiffness (1 item), pain (4 items), and functions of daily living (2 items). Scores range from 0 to 100 with a score of 0 indicating total knee disability and 100 indicating perfect knee health.
EQ-5D-5L | 12 months
  The change in measured EQ-5D-5L scale from baseline. This outcome instrument is composed of five sub-scales containing five questions each. The point range for each sub-scale is from 1 to 5, with "1" indicating the best study subject condition and "5" indicating the worst study subject condition. Thus, the minimum and maximum scores per sub-scale are 1 and 5, respectively, and such scores for the entire instrument are 5 (best study subject condition) and 25 (worst study subject condition). The sub-scale topics are: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression
Global Perceived Effect (GPE) | 12 months
  The measured Global Perceived Effect scale. The Global Perceived Effect is a 7-point scale: 1 point = "worst ever", 2 points = "much worse", 3 points = "worse", 4 points = "not improved but not worse", 5 points = "improved", 6 points = "much improved", 7 points = "best ever". There are no sub-scales.

OTHER OUTCOMES:
Numeric Rating Scale (NRS) | 24 months
  The proportion of subjects whose knee pain is reduced by ≥ 50% based on the NRS. The NRS is an 11-point scale (0 points to 10 points), where 0 points equals "no pain" and 10 points equals "worst pain". There are no sub-scales.
Additional Interventions | 24 months
  The proportion of subjects requiring additional intervention for their OA knee pain.
Knee injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS, JR) | 24 months
  The change in KOOS JR score from baseline. The KOOS JR is a short form of the KOOS that assesses patient stiffness (1 item), pain (4 items), and functions of daily living (2 items). Scores range from 0 to 100 with a score of 0 indicating total knee disability and 100 indicating perfect knee health.
EQ-5D-5L | 24 months
  The change in measured EQ-5D-5L scale from baseline. This outcome instrument is composed of five sub-scales containing five questions each. The point range for each sub-scale is from 1 to 5, with "1" indicating the best study subject condition and "5" indicating the worst study subject condition. Thus, the minimum and maximum scores per sub-scale are 1 and 5, respectively, and such scores for the entire instrument are 5 (best study subject condition) and 25 (worst study subject condition). The sub-scale topics are: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression
Global Perceived Effect (GPE) | 24 months
  The measured Global Perceived Effect scale. The Global Perceived Effect is a 7-point scale: 1 point = "worst ever", 2 points = "much worse", 3 points = "worse", 4 points = "not improved but not worse", 5 points = "improved", 6 points = "much improved", 7 points = "best ever". There are no sub-scales.

CONTACTS AND LOCATIONS:
Overall Officials: David Kennedy, MD, Principal Investigator — Vanderbilt Stallworth Rehabilitation Hospital
Locations (7):
- United States (7):
  - University Orthopedics Center, Altoona, Pennsylvania
  - Pain Diagnostics and Interventional Care, Sewickley, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania
  - Piedmont Comprehensive Pain Management, Anderson, South Carolina
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - The Spine and Nerve Centers of St. Francis Hosptial, Charleston, West Virginia